CLINICAL TRIAL: NCT01347567
Title: HF Outpatient Monitoring Evaluation (HOME) Study
Brief Title: Heart Failure (HF) Outpatient Monitoring Evaluation (HOME) Study
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alere San Diego (Industry)
Responsible Party: Sponsor
Organization: Abbott RDx Cardiometabolic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSTE-0135
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure; Systolic Heart Failure; Acute Decompensated Heart Failure
Keywords: Fingerstick BNP test; Home Health Management System; Acute Decompensated Heart Failure; Hospital Readmission; Prevention
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- BNP + Health Management (Experimental): Subjects will provide information from home regarding weight,signs and symptoms, and will perform BNP self testing. This information including BNP results will be used by the investigator as an aid to treatment decisions. BNP results are blinded to subjects.
  Interventions: Other: Interventions with heart failure medications
- Health Management (Active Comparator): Subjects will provide information from home regarding weight, signs and symptoms, and will perform BNP self testing . BNP results will be blinded to the investigator and subject; weight, signs and symptoms will be used by the investigator as an aid to treatment decisions
  Interventions: Other: Interventions with heart failure medications
- Control (Placebo Comparator): Subject will provide information from home regarding weight, signs and symptoms and will perform BNP self testing. All these data will be blinded to the investigator. BNP results will be blinded to the subject.
  Interventions: Other: Interventions with heart failure medications

INTERVENTIONS:
Other: Interventions with heart failure medications — Therapeutic interventions with heart failure medications per decision of treating physician for subjects in all study arms but using the different information available in each study arm.

SUMMARY:
The purpose of this study is to determine if heart failure subjects whose treatment is assisted by home BNP measurements integrated into a home health management system will have better clinical outcomes than subjects whose treatment includes home health management without BNP or than subjects treated by standard care.

DETAILED DESCRIPTION:
Systolic dysfunction heart failure subjects with low ejection fraction and elevated BNP levels admitted to hospital or treated as outpatient for decompensated Heart Failure (HF) are at hight risk for recurrent decompensation and readmission. The objective of this study is to investigate if these patients may benefit from enhanced home monitoring of their HF status.

In the 3 study arms (BNP, Health Management and control groups) home fingerstick BNP levels will be obtained so that frequent data points are available for analysis of trends and variability. These results will remain blinded to the subjects in all study arms and their care providers in the health management and control arms, the investigator and staff will have access to the BNP results only for subjects in the BNP arm and will use this information to aid in therapy decisions.

Subjects are monitored for 180 days as this time period is likely sufficient to differentiate normal biological variation in BNP changes due to impending decompensation.

Patients will be assessed at Day 30,90 and 180 after randomization HF status, patient clinical outcome and treatment adjustments are recorded.

Follow-up telephone calls to subjects at 3 and 6 months after completion of home testing will be conducted in order to determine the possible long-term benefit of home health management with daily BNP testing.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years of age and <75 years of age); AND
2. Admitted to the hospital or treated in an outpatient clinic with a diagnosis of decompensated HF for which treatment will be administered;

i. BNP > 300 pg/mL (or NT-pro-BNP > 1500 pg/mL) during hospital admission or clinic visit.

OR c. Seen in an outpatient setting (i.e. heart failure clinic, general practice or cardiology office, urgent care unit) with a documented history of HF and with signs of worsening HF condition or decompensation, where worsening HF condition is defined as one or more of the following;

i. Increase in NYHA class with worsening symptoms (i.e. dyspnea, fatigue) at same level of activity ii. Symptoms requiring change in dosage of one or more of the following medications:

1. diuretic
2. beta blocker
3. ACE inhibitor iii. Physical evaluation consistent with worsening HF signs (i.e. elevated JVP, ankle edema, dyspnea, abdominal distension, >4 lb or >1.8 kg weight increase in past week) iv. HF admission in last 30 days with a documented BNP > 300 pg/mL (or NT-pro-BNP > 1500 pg/mL) during or since admission AND d. Presence of left ventricular systolic dysfunction (ejection fraction <40%); e. Successfully trained and deemed proficient on how to perform a fingerstick and to use the Test System. Each subject will undergo two proficiency assessments.

   i. The first assessment will be performed at the time in which the subject is found to meet the inclusion criteria, and deemed willing, able and reliable to complete the study tasks, and following initial training on the use of the test system. Successful completion of this first proficiency assessment will result in the enrolment of the subject into the study.

   The second assessment will be performed following one week (7 days ± 2 days) of home testing to demonstrate retention of the training. Successful completion of this second proficiency assessment will result in randomization of the subject into one of the three study arms of the study. Failure to demonstrate proficiency at this second assessment will result in the withdrawal of the subject from the study.

   Exclusion criteria:
   1. Unwilling or unable to provide written informed consent;
   2. Acute coronary syndrome (ACS) that is a primary diagnosis; or secondary diagnosis that is concomitant with the primary diagnosis of decompensated HF and for which treatment will be provided.

      Note: A history of ACS is not cause for exclusion if it is not concomitant with the present decompensated HF for which admission is being made. Small elevations in cardiac troponin that are considered by the treating physician to be associated with myocardial injury due to the acute decompensated HF and not due to a concomitant ACS or myocardial infarction are not a basis for exclusion.
   3. Previous cardiac transplantation - or cardiac transplantation anticipated within 3 months;
   4. Current or planned use of a left ventricular assist device (LVAD), use of outpatient intravenous inotropic HF therapy, major surgical procedure or percutaneous coronary intervention within 3 months;
   5. Life expectancy less than 6 months due to causes other than HF or cardiovascular disease (e.g., cancer);
   6. End stage renal disease (dialysis dependency);
   7. Receiving any investigational medication;
   8. Hematocrit outside the 25 to 50% range of the HeartCheck system;
   9. Prisoner or other institutionalized or vulnerable individual;
   10. Dementia, tremors or other impediments to performing daily home BNP testing via fingerstick (unless BNP testing will be conducted by qualified caregiver);
   11. Deemed by the investigator not to be likely to comply with study-mandated procedures or instructions;
   12. Residence in regions where either transmission of test system data or home visits are not possible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Average number of "hard' events per subject | Over 180 days
  With hard events defined as:
  * HF related death,
  * HF related readmissions to the hospitaL,
  * IV treatment with diuretics or unusual oral diuretic change in ER
  * Unplanned outpatient treatments for decompensated HF

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth McDonald, Professor, Study Director — St Vincent's Private Hospitale Ltd, Dublin, Ireland; Henry Dargie, Professor, Principal Investigator — Western Infirmary, Glasgow, UK; Theresa McDonagh, Professor, Principal Investigator — Royal Brompton, London, UK; John Atherton, Professor, Principal Investigator — Royal Brisbane and Women's Hospital, Herston, Australia; Henry Krum, Professor, Principal Investigator — Monash University; Richard Thoughton, Professor, Principal Investigator — University of Otago, Christchurch, New Zealand; Rob Doughty, Professor, Principal Investigator — University of Auckland, Victoria, New Zealand; Faiez Zannad, Professor, Principal Investigator — Institut Lorrain du Coeur et des Vaisseaux, CHU Nancy, Vandoeuvre-les-Nancy, France; Ulf Dahlstrom, Professor, Principal Investigator — Linkoping University Hospital, Sweden; P Van der Meer, Doctor, Principal Investigator — University Medical Center Groningen, the Netherlands; Franz Kleber, Professor, Principal Investigator — Klinikum Ernst von Bergmann, Akademisches Lehrankenhaus der Charite Universitätsmedizin Berlin, Germany
Locations (7):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia
- St Vincent's Private Hospitale LTd, Dublin, Ireland
- University Medical Center Groningen, Gronongen, Netherlands
- New Zealand (2):
  - University of Auckland, Auckland
  - Department of Medicine, University of Otago, Christchurch
- Linkoping University Hospital, Linköping, Sweden
- Royal Brompton Hospital, London, United Kingdom